CLINICAL TRIAL: NCT03117764
Title: The 1-minute-sit-to-stand Test is Practical to Assess and Follow the Muscle Weakness in Cystic Fibrosis.
Brief Title: 1STST and Muscle Weakness in CF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Hardy, MD, Pneumology assistant, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hardy
Record Dates: First submitted 2017-03-31; First posted 2017-04-18 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute IV AB for exacerbation at hospital (Active Comparator): The study will compare muscular strength of hospitalised patients who receive specific exercise training, with patients who follow their antibiotherapy at home without specific exercise training.
  Interventions: microfet dynamometer, 1 minute sit to stand test, accelerometer.
  Interventions: Device: Microfet Dynamometer; Behavioral: 1 minute sit to stand test; Device: Accelerometer
- Acute IV AB for exacerbation at home (Experimental): The study will compare muscular strength of hospitalised patients who receive specific exercise training, with patients who follow their antibiotherapy at home without specific exercise training.
  Interventions: microfet dynamometer, 1 minute sit to stand test, accelerometer.
  Interventions: Device: Microfet Dynamometer; Behavioral: 1 minute sit to stand test; Device: Accelerometer

INTERVENTIONS:
Device: Microfet Dynamometer — To evaluate muscular strength, the investigators will measure quadriceps force at the beginning of the cure and at the end with a functional test, the 1-minute Sit-to-Stand test, and a maximal isometric force test, with the Microfet2dynamometer. Those tests are not invasive and easy to realise.
  The investigators will estimate the physical activity of the patients with an accelerometer that they will each carry 72 hours, during the cure.
  Patients who undergo their cure at the hospital will follow a specific training program with the physiotherapist.
Behavioral: 1 minute sit to stand test — To evaluate muscular strength, the investigators will measure quadriceps force at the beginning of the cure and at the end with a functional test, the 1-minute Sit-to-Stand test, and a maximal isometric force test, with the Microfet2dynamometer. Those tests are not invasive and easy to realise.
  The investigators will estimate the physical activity of the patients with an accelerometer that they will each carry 72 hours, during the cure.
  Patients who undergo their cure at the hospital will follow a specific training program with the physiotherapist.
Device: Accelerometer — To evaluate muscular strength, the investigators will measure quadriceps force at the beginning of the cure and at the end with a functional test, the 1-minute Sit-to-Stand test, and a maximal isometric force test, with the Microfet2dynamometer. Those tests are not invasive and easy to realise.
  The investigators will estimate the physical activity of the patients with an accelerometer that they will each carry 72 hours, during the cure.
  Patients who undergo their cure at the hospital will follow a specific training program with the physiotherapist.

SUMMARY:
The investigators know that peripheral muscle weakness and exercise intolerance are prevalent (56%) in cystic fibrosis (Trooster et al, 2009). Physical inactivity is likely to be an important underlying factor. Those conditions are associated with a poor prognosis (Nixon et al, 1992). The effect of intravenous antibiotherapy on peripheral muscle and physical activity remains unclear.

The aim of the study is to evaluate the impact of intravenous antibiotherapy on peripheral muscular strength in patients with cystic fibrosis (adults and children) who receive intravenous antibiotherapy for an acute exacerbation or electively (decline in lung function without exacerbation).

DETAILED DESCRIPTION:
Background Peripheral muscle weakness and exercise intolerance are prevalent (56%) in cystic fibrosis (Trooster et al, 2009). Physical inactivity is likely to be an important underlying factor. Those conditions are associated with a poor prognosis (Nixon et al, 1992). The effect of intravenous antibiotherapy on peripheral muscle and physical activity remains unclear. Wieboldt et al showed that quadriceps strength at the hospital admission for an exacerbation was lower than before and one month after hospitalisation while Burtin et al showed that individual changes in quadriceps force were correlated with daily time spent activities of at least moderate intensity (Wieboldt et al, 2012; Burtin et al, 2013). The effect of intravenous antibiotherapy itself is poorly known in cystic fibrosis. Moreover, they did not study the impact on muscular strength of hospitalisation versus home treatment. In contrast, in COPD, it is well known that exacerbations are associated with a decline of muscle mass and strength and that repeated exacerbations lead to a more rapid decrease in fat free mass (Spruit et al, 2003; Jones et al, 2015; Joppa et al, 2016).

Hypothesis We think that exacerbations aggravate factors underlying muscle weakness as physical inactivity, systemic inflammation and anabolic status. Moreover, hospitalisation itself might be a reason of inactivity as patients spent all the day inside their room compared to patients who follow their treatment at home and continue their usual life.

Aim The aim of our study is to evaluate the impact of an intravenous antibiotherapy on peripheral muscular strength in patients with cystic fibrosis.

Methods We would compare patients (adults and children) who receive intravenous antibiotherapy for an acute exacerbation, with patients who receive elective intravenous antibiotherapy (decline in lung function without exacerbation). We will also compare hospitalised patients who receive specific exercise training, with patients who follow their antibiotherapy at home without specific exercise training. We will have a stable patients group as control. To evaluate muscular strength we plan to measure quadriceps force at the beginning of the cure and at the end with a functional test, the 1-minute Sit-to-Stand test and a strength (isometric) test, with the Microfet2dynamometer. Those test are not invasive, easy to realise and have already been used in other studies (Ozalevli, 2005). We will quantify the physical activity level of the patients with an accelerometer that they will carry during 72 hours, during the first week of the treatment.

ELIGIBILITY:
Inclusion Criteria:

- patients with cystic fibrosis following the definition of Rosentein et al (1997), who undergo an intravenous antibiotic cure for an acute exacerbation or electively since we notice a decline of respiratory lung function

Exclusion Criteria:

* orthopaedic conditions interfering with mobility or the assessment of skeletal muscle force,
* a pregnancy,
* a pulmonary graft
* a negative response for the informed consent.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change from peripheral muscular strength at 14 days. | At day 0 and day 14 of IV AB
  To evaluate the impact of intravenous antibiotherapy on peripheral muscular strength. Is the impact negative or positive?

CONTACTS AND LOCATIONS:
Overall Officials: hardy Sophie, MD, Principal Investigator — St Luc
Locations (1):
- Hardy Sophie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No